CLINICAL TRIAL: NCT02355938
Title: Role of Fidaxomicin in a Patient Population With Problematic Clostridium Difficile Infection
Brief Title: Use Of Oral Fidaxomicin Vs. Oral Vancomycin For Clostridium Difficile Infection In Patients With Spinal Cord Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost funding due to low enrollment.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Rabih Darouiche, Medical Doctor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIS-000116; H-32358 (Other: Baylor College of Medicine)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Clostridium Difficile; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Fidaxomicin; Cellulose; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fidaxomicin Arm (Experimental): Oral Fidaxomicin 200 mg every 12 hours (Placebo for 2 doses) for 10 days
  Interventions: Drug: Fidaxomicin 200 mg; Drug: Placebo
- Vancomycin Arm (Active Comparator): Oral Vancomycin 125 mg every 6 hours for 10 days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Fidaxomicin 200 mg — Fidaxomicin 200 mg every 12 hours
  Other Names: Dificid
  Arms: Fidaxomicin Arm
Drug: Placebo — 1 dose of placebo every 6 hours x 2 doses
  Other Names: Cellulose Capsule
  Arms: Fidaxomicin Arm
Drug: Vancomycin — Vancomycin 125 mg every 6 hours
  Other Names: Vancocin
  Arms: Vancomycin Arm

SUMMARY:
The primary purpose of this study is to compare the clinical outcomes of cure and recurrence of Clostridium difficile infection in spinal cord injured patients who are treated with oral Fidaxomicin vs. oral Vancomycin. The secondary aim of this study is to compare the overall costs of treatment of Clostridium difficile infection in the two study groups.

DETAILED DESCRIPTION:
In recent clinical trials, comparing oral Vancomycin versus oral Fidaxomicin to treat Clostridium difficile, oral Fidaxomicin was shown to be the same in effectiveness as oral Vancomycin, but showed a decrease in recurrence of Clostridium difficile by ten percentage points. Based on experience with patients in our 40-bed spinal cord injury unit at the Michael E. DeBakey VA Medical Center (MEDVAMC), Clostridium difficile infection is more problematic in patients with spinal cord injury than in the general hospitalized patient population. Compared to the general population of hospitalized patients, patients with spinal cord injury are more likely to have: (1) a higher transmission of Clostridium difficile from one patient to another often via the health care worker due to their having a neurogenic bowel (2) a longer and more complicated course of Clostridium difficile infection-associated diarrhea since neurogenic bladder may delay excretion of toxins and predispose to bowel accidents; and (3) a higher overall cost of treatment in terms of extended hospitalization (most patients with spinal cord injury who suffer from Clostridium difficile infection do not get discharged from the hospital until the symptoms of course of Clostridium difficile infection are resolved. Fidaxomicin is the first in a new class of narrow spectrum macrocyclic antibiotic drugs. It is a non-systemic, meaning it is minimally absorbed into the bloodstream, and it is bactericidal, meaning it attacks and kills the bacteria it comes in contact with. It has demonstrated selective eradication of pathogenic Clostridium difficile with minimal disruption to the numerous species of bacteria that make up the normal, healthy intestinal flora. The maintenance of normal physiological conditions in the colon can reduce the probability of recurrence of a Clostridium difficile infection. Since clearance of Clostridium difficile infections is problematic in the spinal cord injured patients, this antimicrobial agent may show a trend for clinical superiority and a reduction in recurrence of infection within the spinal cord injury population resulting in a shorter hospital stays and reduced costs.

ELIGIBILITY:
Inclusion Criteria:

* Ability of subject to provide an informed consent
* Legally Authorized Representative-Adult must provide consent in case the subject is unable to consent
* Diagnosis of Clostridium difficile disease based on clinical manifestations (change in bowel habits, at least 2 more unformed bowel movements as compared to baseline neurogenic bowel function in the same patient in the 24-hour period prior to randomization)
* Lab data (positive polymerase chain reaction test for Clostridium difficile in a stool specimen obtained within 72 hours before randomization)
* Patient has not received antibiotics that are active against Clostridium difficile for any more than 24 hours prior to being screened for this study.

Exclusion Criteria:

* Receipt of agents (oral Vancomycin, oral or IV Metronidazole, oral rifamdin, oral bacitracin, or oral fusidic acid) that are active against Clostridium difficile for longer than 24 hours after randomization
* Life-threatening or fulminant Clostridium difficile infection, presence of toxic megacolon, and history of inflammatory bowel disease (Crohn's disease and ulcerative colitis)
* Allergy to study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cure of Clostridium Difficile | 10 Days
  Decrease in number and frequency of loose stools

SECONDARY OUTCOMES:
Cost Benefit Analysis | Hospitalization cost 6 months before and 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Enrollment to low for statistical analysis.